CLINICAL TRIAL: NCT06615921
Title: A Multi-country, Multi-center, Retrospective Chart Review to Describe the Use of Maribavir and Its Effectiveness in Patients With Post-Transplant Cytomegalovirus Infection/Disease
Brief Title: A Study of Maribavir in Adults With Post-transplant Cytomegalovirus (CMV) Infection
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-620-5010
Record Dates: First submitted 2024-08-23; First posted 2024-09-27 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Cytomegalovirus (CMV)
Keywords: Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants With CMV Infection Refractory: Participants who had a CMV infection/disease that is refractory to treatment (with or without resistance). Data will be retrospectively collected from date of solid organ transplant (SOT) or hematopoietic stem cell transplant (HSCT) up to the start date of chart abstraction, death or loss to follow-up, whichever comes first. Participants will be considered as refractory if they show no change or increased viremia after at least 2 weeks of appropriately dosed antiviral therapy.
  Interventions: Other: No Intervention
- Participants With CMV Infection Intolerant: Participants with CMV infection intolerant to anti-CMV treatment. Data will be retrospectively collected from date of SOT/HSCT up to the start date of chart abstraction, death or loss to follow-up, whichever comes first. Intolerant participants identified based on physician judgment.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The main aim of this study is to check how effective the treatment with Maribavir has been to remove the CMV viruses from the blood of an adult person with CMV infection after a transplant. Other aims are to learn more about how maribavir is used in normal clinical routine, study the profiles of adults treated with maribavir, and what other treatments have been given, and describe healthcare resources used for CMV management.

Only data already available in the medical records of the participants will be reviewed and collected during this study.

DETAILED DESCRIPTION:
This study will include two main periods of retrospective data collection from medical charts: the pre-index period and the post-index period. The index date is defined as the date of initiation of maribavir dosing, as documented in the medical records. The pre-index period covers the time from the transplant date to the index event, while the post-index period starts at the index event and ends at the date of chart abstraction, death, or loss to follow-up, whichever comes first.

ELIGIBILITY:
Inclusion criteria:

* Aged greater than or equal to (>=) 18 years at the time of consent or start of chart abstraction in case a consent waiver will be allowed as per local regulation.
* Received an HSCT/SOT.
* Diagnosed with CMV infection/disease any time after the HSCT/SOT date.
* Initiated maribavir at least 4 months before the chart abstraction date (or at time of Central Ethics Committee [CEC]/Local Ethics Committee [LEC] submission as per local regulation).
* Participants with hospital medical chart available, who signed an informed consent form before starting any study procedures (unless waiver is allowed as per local regulation).

Exclusion criteria:

* Participants who do not provide informed consent, where consent is required per country regulations.
* Participants who participated to Clinical Trials investigating maribavir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have been diagnosed with Post-Transplant Cytomegalovirus infection/disease in several European countries.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Viremia Clearance Before the End of Maribavir Treatment | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  CMV viremia clearance is defined as a negative Quantitative Polymerase Chain Reaction (PCR) result. A PCR result is defined as negative if CMV DNA is undetectable or below the lower limit of quantification as per local laboratory practice. Number of participants with the last CMV quantitative negative PCR result before the end of maribavir treatment will be reported.

SECONDARY OUTCOMES:
Participants Categorized Based on Demographic Characteristics | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants will be reported by their demographic characteristics (age, sex, past conditions and comorbidities).
Participants Categorized by Transplant-Related Characteristics | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants will be reported by transplant-related characteristics (type of transplant [HSCT/SOT]), transplant indication, donor and recipient CMV serostatus).
Participants Characterized by Previous CMV Infection (Medical History) | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants with prior CMV infections and clinical manifestations of CMV disease before Index CMV episode. Index CMV episode is defined as first CMV episode treated with maribavir.
Participants Characterized by Use of Prior Anti-CMV Treatment Strategies | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants will be reported by treatments used (e.g. valganciclovir, ganciclovir, cidofovir, foscarnet or letermovir), by number and sequence of treatments/per CMV episode, by treatment strategy (e.g. prophylaxis, pre-emptive, treatment) before Index CMV episode. Index CMV episode is defined as first CMV episode treated with maribavir.
Duration of Each Treatment With Maribavir During Index and/or Post-Index CMV Episodes | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Duration between start and end of treatment during Index and Post-index CMV episodes will be reported. Index CMV episode is defined as first CMV episode treated with maribavir. Post-index CMV episode is defined as first CMV recurrent episode after Index episode.
Number of Repeated Treatments With Maribavir During Index and/or Post-Index CMV Episodes | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of repeated treatments with maribavir per CMV episode will be reported during index and/or post-index CMV episodes.
Maribavir Administration by Line of Therapy During Index and/or Post-Index CMV Episodes | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants who received maribavir, as derived from the treatments sequence within a specific CMV episode, stratified by line of therapy.
Participants With Maribavir Dose Adjustments During Index and/or Post-Index CMV Episodes | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants with maribavir dose adjustments and average dose adjustments will be reported.
CMV Viral Load Prior to Maribavir Initiation, During Treatment With Maribavir, and After Discontinuation | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Available CMV viral loads of interest prior to maribavir initiation, during treatment with maribavir, and after discontinuation will be reported for each maribavir treatment administered.
Reasons for Initiating and Discontinuing Maribavir Treatment During Index and/or Post-Index CMV Episodes | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants categorized by their reasons for initiating and discontinuing maribavir treatment will be reported.
Place of Initiation of Maribavir Treatment | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants categorized by place of initiation of maribavir treatment (Home/Hospital) will be reported.
Duration of Maribavir Treatment During Hospital In-patient Stay | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of days of maribavir treatment during hospital in-patient stay will be reported.
Participants who Received Maribavir Monotherapy or Maribavir in Combination With Other Antivirals | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants who received maribavir as monotherapy or in combination with other antivirals such as valganciclovir, ganciclovir, letermovir, cidofovir or foscarnet will be reported.
Participants who Received Concomitant Use of CMV-Specific IgG During Index and/or Post-Index CMV Episodes | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants who received concomitant use of CMV-specific IgG during maribavir treatment will be reported.
Participants With Concomitant Use of Granulocyte Colony-Stimulating Factor (G-CSF) | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants who received concomitant use of G-CSF during maribavir treatment will be reported.
Participants With Immunosuppressive Therapy Adjustments During Index and/or Post-Index CMV Episodes | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants with immunosuppressive therapy adjustments during Index and/or Post-index CMV episodes will be reported.
Time to First CMV Viremia Clearance After Initiation of Maribavir During Index and/or Post-Index CMV Episodes | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Time to first CMV viremia clearance (first negative PCR) after initiation of maribavir will be reported. CMV viremia clearance is defined as a negative Quantitative PCR result. A PCR result is defined as negative if CMV DNA is undetectable or below the lower limit of quantification as per local laboratory practice.
Time to First CMV Viremia Control After Initiation of Maribavir During Index and/or Post-Index CMV Episodes | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Time to first CMV viremia control after initiation of maribavir will be reported. Viremia control is defined as at least a 1 log10 decrease in CMV DNA levels in blood, serum, or plasma, assessed through PCR, from the peak viral load before initiation of maribavir treatment and peak viral load at subsequent weeks of maribavir treatment.
Participants With CMV Viremia Control per Week After Initiation of Maribavir During Index and/or Post-Index CMV Episodes | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants with CMV viremia control per week after initiation of maribavir will be reported. Viremia control is defined as at least a 1 log10 decrease in CMV DNA levels in blood, serum, or plasma, assessed through PCR, from the peak viral load before initiation of maribavir treatment and peak viral load at subsequent weeks of maribavir treatment.
Participants With Cumulative CMV Viremia Control at the End of Maribavir Treatment During Index and/or Post-Index CMV Episodes | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants with cumulative CMV viremia control at the end of maribavir treatment will be reported. Viremia control is defined as at least a 1 log10 decrease in CMV DNA levels in blood, serum, or plasma, assessed through PCR, from the peak viral load before initiation of maribavir treatment and peak viral load at subsequent weeks of maribavir treatment.
Incidence of Tissue Invasive Disease During Index and/or Post-Index CMV Episodes | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Percentage of participants with tissue invasive disease during Index and/or Post-index CMV episodes will be reported.
Time to Tissue Invasive Disease During Index and/or Post-Index CMV Episodes | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Time to event of tissue invasive disease will be reported.
Incidence of CMV Syndrome Disease During Index and/or Post-Index CMV Episodes | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Percentage of participants with CMV syndrome disease will be reported.
Time to CMV Syndrome Disease During Index and/or Post-Index CMV Episodes | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Time to event of CMV syndrome disease will be reported.
Participants With Reduction or Resolution of CMV Disease/Syndrome at the End of Maribavir Treatment | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants with reduction or resolution of CMV disease/syndrome at the end of maribavir treatment will be reported.
Time to Reduction or Resolution of CMV Disease/Syndrome After Maribavir Initiation | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Time to reduction or resolution of CMV disease/syndrome after maribavir initiation will be reported.
Participants With Recurrent CMV Viremia (Post-Index CMV Episode) | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants with asymptomatic and symptomatic recurrent CMV viremia (Post-index CMV episode) will be reported.
Time From Maribavir Discontinuation to Next CMV Treatment and Anti-CMV Agent Used | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Time from maribavir discontinuation to next CMV treatment and anti-CMV agent will be reported.
Participants With Anti-CMV Detected Resistance Mutations in the Study Population | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants with detected anti-CMV resistance mutations prior to and after initiation of maribavir will be reported.
Participants With Anti-CMV Treatment Related Adverse Events of Special Interest (AESI) | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants with Anti-CMV Treatment Related AESI will be reported. AESI will include myelosuppression (for example, leucopenia, thrombocytopenia, lymphopenia, neutropenia, etc.), nephrotoxicity and taste disturbances.
Participants With Abnormal Laboratory Parameters Related to AESI | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants with abnormal laboratory parameters related to AESI will be reported. Laboratory parameters refer to complete blood count, glomerular filtration, etc.
Participants With AESI Related to the Administration of Maribavir | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants with AESI related to the administration of maribavir will be reported.
Participants With Outpatient Visit/Hospitalization Related to CMV Management | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Number of participants with outpatient visit/hospitalization related to CMV management will be reported. Participants will be categorized by type of visit (outpatient, hospitalizations/emergency department visits), primary reason for the visit, CMV-related exams/procedures.
Length of Hospital Stay in Days for CMV-related Hospitalizations | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Length of hospital stay in days for CMV -related hospitalizations will be reported.
Duration in Days of Critical Care against Non-critical Care | From transplantation date until start of chart abstraction or date of death from any cause, whichever comes first, up to approximately 32 months
  Duration in days of stay in critical care and non-critical care will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (45):
- Medical University of Vienna Dept. of Nephrology and Dialysis, Vienna, Austria
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark
- France (10):
  - Groupe Hospitalier Pellegrin - CHU BORDEAUX, Bordeaux
  - Department of Nephrology, University Hospital of Dijon, Dijon
  - Hopital Claude Huriez CHRU Lille, Lille
  - CHU Montpellier, Montpellier
  - CHU De Nice Hopital Pasteur 2, Nice
  - Hopital Saint-Louis AP-HP Pitor, Paris
  - APHP, Sorbonne University, Pitie Salpetriere Hospital, Paris
  - Necker-Enfants Malades Hospital, Paris
  - Hopitaux Universitaires de Strasbourg, Strasbourg
  - Toulouse University Hospital - Hopital de Rangueil, Toulouse
- Germany (11):
  - Uniklinik RWTH Aachen, Aachen
  - Charite, Dept of Nephrology, Berlin
  - Clinic for Infectiology - Essen, Essen
  - University Hospital Greifswald, Greifswald
  - Clinic for stem cell transplantation - Hamburg (UKE), Hamburg
  - Hannover Medical School - Resp Medicine, Hanover
  - Uniklinik Leipzig, Leipzig
  - Medicine Clinic of Johannes Gutenberg - Mainz university, Mainz
  - Ludwig-Maximilians University (LMU) Hospital, Munich
  - University of Ulm, Ulm
  - Universitaetsklinikum Wuerzburg, Würzburg
- Policlinico Gemelli - Roma, Roma, Italy
- Netherlands (2):
  - Erasmus MC Cancer Institute, Rotterdam
  - UMC Utrecht (Hematology), Utrecht
- Serbia (2):
  - University of Belgrade, Belgrade
  - Clinical Center of Vojvodina, Novi Sad
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de Cruces, Bilbao
  - Hospital Virgen de las Nieves, Granada
  - Hospital Dr. Negrin, Las Palmas
  - Hospital 12 de Octubre, Madrid
  - Hospital Puerta del Hierro, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
- University Hospital of Geneva, Geneva, Switzerland
- United Kingdom (9):
  - University Hospitals Birmingham, Birmingham
  - Royal Papworth Hospital (Cambridge), Cambridge
  - University College Hospital London, London
  - Kings College Hospital (London), London
  - Royal Marsden Hospital (London), London
  - Manchester Royal Infirmary, Manchester
  - Freeman Hospital Newcastle upon Tyne, Newcastle
  - Nottingham University Hospital NHS trust (Queens Medical Centre), Nottingham
  - University Hospital Southampton NHS FT, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/23f41f1b0bb64428??page=1&idFilter=TAK-620-5010